CLINICAL TRIAL: NCT00987415
Title: Xanthine Oxidase Inhibition for Hyperuricemic Heart Failure Patients
Brief Title: Using Allopurinol to Relieve Symptoms in Patients With Heart Failure and High Uric Acid Levels
Acronym: EXACT-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00020011; 5U10HL084904 (NIH)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Heart Failure; Elevated Serum Uric Acid
MeSH Terms: conditions — Heart Failure | interventions — Allopurinol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allopurinol (Active Comparator): Allopurinol 300 mg daily for one week, then 600 mg daily to complete 24 weeks.
  Interventions: Drug: allopurinol
- sugar pill (Placebo Comparator): Matching placebo 300 mg daily for one week, then 600 mg daily to complete 24 weeks.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: allopurinol — Allopurinol 300 mg daily for one week, then 600 mg daily to complete 24 weeks.
  Arms: allopurinol
Drug: sugar pill — Matching placebo 300 mg daily for one week, then 600 mg daily to complete 24 weeks.
  Arms: sugar pill

SUMMARY:
The purpose of this study is to determine whether allopurinol is effective in relieving symptoms of patients with heart failure and high blood uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class II-IV heart failure due to ischemic or non-ischemic cardiomyopathy.
* Left ventricular ejection fraction ≤ 40% by echocardiography- Heart failure symptoms for 3 months despite standard treatment.
* Serum uric acid level ≥ 9.5 mg/dl.
* At least one of the following additional markers of increased risk: Hospitalization, ER visit or urgent clinic visit for heart failure requiring IV diuretics within the previous 12 months; Left ventricular ejection fraction ≤ 25; B-type natriuretic peptide level > 250 pg/ml

Exclusion Criteria:

* Hypertrophic or restrictive cardiomyopathy, constrictive pericarditis, biopsy-proven myocarditis, severe stenotic valvular disease, or complex congenital heart disease.
* Acute coronary syndrome, PCI or CABG within 3 months.
* Current ventricular assist device or ventricular assist device or heart transplant likely within the next 6 months.
* Uncontrolled hypertension (i.e., SBP > 170 mm Hg or DBP > 110 mm Hg)
* Serum creatinine > 3 mg/dL or estimated GFR < 20 ml/min.
* Evidence of active hepatitis with ALT and AST greater than 3x normal.
* Any condition other than HF which could limit the ability to perform a 6-minute walk test
* Any diseases other than HF which are likely to alter the patient's global perception of status or quality of life over a period of 6 months.
* Receiving treatment with allopurinol currently or within 30 days, or having symptomatic hyperuricemia which requires treatment with allopurinol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Braunwald, MD, Study Chair — Harvard University; Alice Mascette, MD, Study Director — National Heart, Lung, and Blood Institute (NHLBI); Adrian Hernandez, MD, Principal Investigator — Duke University
Locations (10):
- United States (9):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Harvard University, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals-Case Medical Center, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Univ. of Utah Health Sciences Center, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
- University of Montreal, Montreal PQ, Canada

REFERENCES:
- [Derived] Givertz MM, Anstrom KJ, Redfield MM, Deswal A, Haddad H, Butler J, Tang WH, Dunlap ME, LeWinter MM, Mann DL, Felker GM, O'Connor CM, Goldsmith SR, Ofili EO, Saltzberg MT, Margulies KB, Cappola TP, Konstam MA, Semigran MJ, McNulty SE, Lee KL, Shah MR, Hernandez AF; NHLBI Heart Failure Clinical Research Network. Effects of Xanthine Oxidase Inhibition in Hyperuricemic Heart Failure Patients: The Xanthine Oxidase Inhibition for Hyperuricemic Heart Failure Patients (EXACT-HF) Study. Circulation. 2015 May 19;131(20):1763-71. doi: 10.1161/CIRCULATIONAHA.114.014536. Epub 2015 Apr 14. PMID 25986447
- [Derived] Fravel MA, Ernst ME. Management of gout in the older adult. Am J Geriatr Pharmacother. 2011 Oct;9(5):271-85. doi: 10.1016/j.amjopharm.2011.07.004. Epub 2011 Aug 17. PMID 21849262
- See also: Trial Website — http://www.hfnetwork.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allopurinol | Sugar Pill
Started | 128 | 125
Completed | 119 | 116
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Sugar Pill | Total
Number analyzed (Participants) | 128 | 125 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (14.2) | 61.8 (13.1) | 61.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 110 | 98 | 208
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 42 | 74
  White | 91 | 78 | 169
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 126 | 124 | 250
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 92 | 92 | 184
  Canada | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: A Composite Clinical Endpoint (CCE) That Classifies Subject's Clinical Status as Improved, Worsened, or Unchanged.
Description: CCE composed of 3-level categorical variable with options that include worsened, unchanged or improved
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Allopurinol | Sugar Pill
Number analyzed (Participants) | 128 | 125
participants
  Worsened | 58 | 58
  Unchanged | 54 | 43
  Improved | 16 | 24

2. Secondary Outcome: Change in Quality of Life (KCCQ).
Description: Kansas City Cardiomyopathy (KCCQ) overall summary score - The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline to 12 weeks
Population: Participants analyzed included those patients who had complete data for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allopurinol | Sugar Pill
Number analyzed (Participants) | 120 | 112
units on a scale | 4.45 (15.42) | 3.38 (19.43)

3. Secondary Outcome: Change in Submaximal Exercise Capacity (6-MWT)
Description: 6-Minute Walk Test
Time Frame: Baseline to 12 weeks
Population: Participants analyzed included those patients who had complete data for this endpoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Allopurinol | Sugar Pill
Number analyzed (Participants) | 107 | 104
meters | 9.5 (77.2) | 9.5 (83.5)

4. Secondary Outcome: Change in Quality of Life (KCCQ)
Description: as for outcome 2
Time Frame: Baseline to 24 weeks
Population: Participants analyzed included those patients who had complete data for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allopurinol | Sugar Pill
Number analyzed (Participants) | 118 | 111
units on a scale | 1.13 (18.89) | 4.68 (21.02)

5. Secondary Outcome: Change in Submaximal Exercise Capacity (6-MWT)
Description: 6-Minute Walk Test
Time Frame: Baseline to 24 weeks
Population: Participants analyzed included those patients who had complete data for this endpoint.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Allopurinol | Sugar Pill
Number analyzed (Participants) | 108 | 94
meters | 18.1 (86.4) | 20.7 (86.0)

ADVERSE EVENTS:
Arm/Group | Allopurinol | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 25/128 | 19/125
Other Adverse Events (participants affected / at risk) | 88/128 | 64/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol (N=128) | Sugar Pill (N=125)
Upper Gastrointestinal Hemorhage (Gastrointestinal disorders) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 4 | 1
Anticoagulation Drug Level above Therapeutic (Investigations) | 2 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diarhea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 0 | 1
Diabeties Mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol (N=128) | Sugar Pill (N=125)
Abdominal discomfort (Gastrointestinal disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Blood creatinine increased (Investigations) | 1 | 3
Gout (Metabolism and nutrition disorders) | 9 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Headache (Nervous system disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 11 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No